CLINICAL TRIAL: NCT03818165
Title: Phase 1b Study of the Efficacy and Safety of CAR2 Anti-CEA CAR-T Cell Hepatic Infusions for Pancreatic Carcinoma Patients With CEA+ Liver Metastases Resistant to Standard Therapy Using the HITM Method and Pressure Enabled Delivery Device
Brief Title: Phase 1b Study of CAR2Anti-CEA CAR-T Cell Hepatic Infusions for Pancreatic Carcinoma Patients With CEA+ Liver Metastases
Acronym: AntiCEA_CART
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Limited enrollment.
Sponsor: Sorrento Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SOR-CART-CEA-001
Record Dates: First submitted 2019-01-23; First posted 2019-01-28 (Actual); Last update posted 2023-01-17 (Actual); Status verified 2023-01

CONDITIONS: Metastatic Pancreatic Carcinoma
Keywords: pancreatic carcinoma; Cacinomaembryonic antigen postive (CEA +); liver metastases; pancreatic cancer; CEA; metastatic pancreatic carcinoma; metastatic pancreatic cancer; phase 1
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Intervention Model Description: Three doses of CAR2 Anti-CEA CAR T Cells 1 x 10e10 cells by hepatic artery infusion (on Days 1, 8, and 15) of each 28-day cycle in the Treatment Period using the HITM method and Surefire device, with IL-2 systemic infusion. Patient may receive up to three 28-day cycles of CAR-T therapy in the Treatment Period.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- CAR2 Anti-CEA CAR-T cell (Experimental): 3 doses of CAR2 Anti-CEA CAR-T cells for each cycle; up to 3 additional cycles received per investigator discretion
  Interventions: Biological: CAR2 Anti-CEA CAR-T cells

INTERVENTIONS:
Biological: CAR2 Anti-CEA CAR-T cells — doses will be delivered by hepatic arterial infusions using pressure enhanced delivery device (PEDD)
  Other Names: Surefire Precision Infusion System; K171355

SUMMARY:
This study is an open-label, single arm phase 1b safety study of CAR2 Anti-CEA CAR-T cell hepatic arterial infusions for pancreatic carcinoma patients with carcinoembryonic antigen positive (CEA+) liver metastases resistant to standard therapy who meet all other eligibility criteria.

DETAILED DESCRIPTION:
Patients will receive weekly 3 doses of CAR2 Anti-CEA CAR-T cells in each 28-day cycle by hepatic arterial infusions using a Pressure Enhanced Delivery Device (PEDD) with low dose systemic IL-2 support. Patients may receive up to 3 cycles of CAR2 Anti-CEA CAR-T cell hepatic arterial infusions, per discretion of the investigator.

All patients who receive investigational CAR-T therapy will be included in the analyses and summaries of safety, efficacy, pharmacokinetic, and pharmacodynamic assessments.

ELIGIBILITY:
Inclusion Criteria:

* Must have documented CEA+ pancreatic adenocarcinoma liver metastases and have failed greater than or equal to 1 line of conventional systemic therapy.
* Must have at least evaluable liver metastases.
* Must have a life-expectancy at least 12 weeks.
* Patients must be willing and able to comply with the study schedule and all other protocol requirements.
* Females of childbearing potential must have 2 negative pregnancy tests, agree to pregnancy tests during the study, and sexually active female and male patients must be willing to use an effective birth control method to avoid pregnancy.

Exclusion Criteria:

* Subjects who have received an investigational study drug within 14 days of leukapheresis or 28 days before receiving first dose of study drug.
* Subjects who have received any approved anticancer medication within 14 days of leukapheresis or 14 days before receiving the first dose of study drug.
* Have any unresolved toxicity greater than Grade 2 from previous anticancer therapy.
* Have a history of confirmed metastases outside the peritoneal cavity, lungs, or liver.
* More than 50% replacement of one or both liver lobes with tumor.
* Has tumor causing biliary obstruction not amenable to stenting.
* Have a high volume of lung or peritoneal metastases.
* Has received any CAR cell line therapies.
* Has any clinically significant low baseline lab results for hemoglobin, platelet counts, and neutrophil counts at screening.
* Has untreated or ongoing intra-abdominal infection or bowel obstruction.
* Has any clinically significant elevated baseline lab results for serum creatinine, AST, and total bilirubin (except for patients in whom hyperbilirubinemia is attributed to Gilbert's syndrome), and alkaline phosphatase at screening regardless of causality.
* Known HIV or acquired immunodeficiency syndrome-related illness, acute or history of chronic hepatitis B or C.
* Female patients who are pregnant or breastfeeding.
* Have active bacterial, viral, or fungal infections.
* Has any significant medical condition, laboratory abnormality, or psychiatric illness that would prevent study participation.
* Left ventricular ejection fraction (LVEF) < 40%.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2019-07-29 (Actual); Primary Completion 2020-01-19 (Actual); Study Completion 2021-05-21 (Actual)

PRIMARY OUTCOMES:
Assess preliminary efficacy by overall survival | 6 months
  As a measure of activity, Overall Survival (OS) will be assessed. The events for the assessment of OS are death events. Time to event endpoints will be estimated using Kaplan-Meier methods. Point estimates and 95% confidence intervals will be provided where applicable.

SECONDARY OUTCOMES:
Assess preliminary efficacy by radiographic response rate using Response Evaluation Criteria in Solid Tumors (RECIST) | 6 months
  As a measure of activity, overall response rate will be assessed by radiographic scans using RECIST criteria. Response will be assessed for each patient over a 6-month timeframe during the treatment and observation phases of the protocol.
Assess preliminary efficacy by metabolic response rate using PET Response Criteria in Solid Tumors (PERCIST) | 6 months
  As a measure of activity, overall response rate will be assessed by radiographic scans using PERCIST criteria. Response will be assessed for each patient over a 6-month timeframe during the treatment and observation phases of the protocol.
Assess preliminary efficacy by response rate using Immune-related Response Criteria (irRC) | 6 months
  As a measure of activity, overall response rate will be assessed by radiographic scans using irRC. Response will be assessed for each patient over a 6-month timeframe during the treatment and observation phases of the protocol.
Assess preliminary efficacy by histologic response rate using pathologic response in biopsy specimens | 6 months
  As a measure of activity, overall response rate will be assessed by pathologic criteria using biopsies of the liver metastases and measuring necrosis and fibrosis. REsponse rates will be assess for each patient over a 6-month timeframe during the treatment and observation phases of the protocol.
Assess preliminary efficacy by serologic response rates by CEA levels | 6 months
  As a measure of activity, overall response rate will be assessed by serologic CEA levels. Response will be assess for each patient over a 6-month timeframe during the treatment and observation phases of the protocol.
Assess preliminary efficacy by serologic response rates by CA 19-9 levels | 6 months
  As a measure of activity, overall response rate will be assessed by serologic CA 19-9 levels. Response will be assess for each patient over a 6-month timeframe during the treatment and observation phases of the protocol.
Assess preliminary efficacy by duration of response in accordance with RECIST criteria | 6 months
  As a measure of activity, duration of response will be measured using radiologic scans and assessed according to RECIST criteria. This will be assess for each patient over a 6-month timeframe during the treatment and observation phases of the protocol.
Assess preliminary efficacy by in-liver progression free survival (PFS) | 6 months
  As a measure of activity, in-liver PFS will be assessed. The events for the assessment of PFS are disease progression and death events. This time to event endpoint will be estimated using Kaplan-Meier methods. Point estimate estimates and 95% confidence intervals will be provided where appropriate.

OTHER OUTCOMES:
Assess if serum cytokine levels correlate with response and/or toxicity to hepatic arterial infusions. | 6 months
  As an exploratory analysis, serum cytokine levels will be measured by ELISA to determine if increases in cytokines predict response and/or toxicity to liver arterial infusions.
Assess if neutrophil:lymphocyte ratios correlate with response | 6 months
  As an exploratory analysis, neutrophil:lymphcyte ratios will be calculated to determine if they correlate with response and/or toxicity.
Assess the persistence of CAR-T cells circulating in blood over time | 6 months
  As an exploratory analysis, circulating CAR-T cells will be analyzed to assess persistence of CAR-T cells during the treatment and observation phases of the study.
Assess the persistence of CAR-T cells in liver tumor biopsies over time | 6 months
  As an exploratory analysis, the engraftment of CAR-T cells in planned liver tumor biopsies will be analyzed to assess persistence of CAR-T cells during the treatment and observation phases of the study.
Assess if circulating tumor cells (CTC) correlate with response | 6 months
  As an exploratory analysis, levels of circulating tumor cells (CTC) will be determined to investigate if decreases in CTC levels correlate with response.

CONTACTS AND LOCATIONS:
Overall Officials: Steven C Katz, MD, Principal Investigator — Roger Williams Medical Center
Locations (1):
- Roger Williams Medical Center, Providence, Rhode Island, United States